CLINICAL TRIAL: NCT04872374
Title: Effects of Parmigiano Reggiano on Exercise Induced Muscle Damage in Older Adults
Brief Title: Effects of Parmigiano Reggiano on Skeletal Muscle Damage in Older Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Padova (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PaRMA.1
Record Dates: First submitted 2021-04-23; First posted 2021-05-04 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-01

CONDITIONS: Old Age; Atrophy; Inflammatory Response; Muscle Soreness
MeSH Terms: conditions — Atrophy; Myalgia | interventions — Whey Proteins

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Young adults (Experimental): participants will perform an eccentric exercise bout after 10 days of dietary supplementation
  Interventions: Dietary Supplement: Parmigiano Reggiano; Dietary Supplement: Whey Protein
- Older adults (Active Comparator): participants will perform an eccentric exercise bout after 10 days of dietary supplementation
  Interventions: Dietary Supplement: Parmigiano Reggiano; Dietary Supplement: Whey Protein

INTERVENTIONS:
Dietary Supplement: Parmigiano Reggiano — subjects will receive 50 g/die of the dietary supplement 10 days before performing the eccentric exercise session
Dietary Supplement: Whey Protein — subjects will receive 20 g/die of the dietary supplement 10 days before performing the eccentric exercise session

SUMMARY:
Aging is associated with the loss of muscle mass and function (sarcopenia) and reduced tissue regenerative capacity.

Eccentric exercise (ECC) is a model of RET that can be used with the elderly, due to the ability of the muscle to combine high muscle strength production with low energy cost. ECC contractions are significantly more damaging to the muscles and produce greater muscle strength, for these reasons there is a greater risk of inducing muscle damage before the muscle is able to adapt.

Parmigiano Reggiano (PR) has some peculiar bromatological characteristics. The proteins contained in it, and in particular the potentially bioactive peptide sequences, can rapidly provide the amino acids necessary to promote muscle growth and repair during exercise. Furthermore, PR can be an important source of fatty acids, of which a significant amount of short-chain fatty acids (SCFA) which are known to have important clinical effects on body composition and metabolic health and can have a systemic anti-inflammatory effect.

Therefore, the central hypothes is that PR consumed during RET can provide more energy substrates and improve muscle recovery. To date, no studies have studied its function on recovery from exercise nor in the elderly.

ELIGIBILITY:
Inclusion Criteria:

* age >60 years old or >18 and < 30 years old
* BMI >18 and <30 kg/m2
* stable body weight in the past 3 months
* valid medical certifacate for practice of physical activity

Exclusion Criteria:

* diabetes or pre-diabetes as for ADA guidelines
* chronic diseases (cardiovascular, liver, respiratory, cancer, etc)
* acute inflammatory status
* regular practice of intense physical activity (>2 sessions/week)
* treatment with steroids in the past 3 months
* regular use of >50g/die of Parmigiano Reggiano

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2021-10-31 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
maximum volountary contraction (MVC) | Change from baseline to up to 5 days
  maximal muscle volountary contraction mesured in Newton

SECONDARY OUTCOMES:
reactive Proteinc C | Change from baseline to up to 5 days
  plasmatic levels of reactive Proteinc C (mg/dL) as a markers of muscle damage
Creatin Kinase | Change from baseline to up to 5 days
  plasmatic levels of Creatin Kinase (mmol/dL) as a markers of muscle damage
IL-6 | Change from baseline to up to 5 days
  plasmatic levels of IL-6 (mg/dL) as a markers of muscle damage
delayed onset muscle soreness (DOMS) | Change from baseline to up to 5 days
  level of delayed onset muscle soreness (DOMS) masured via Visual Analogue Scale (VAS) scale where 0 is the minimal value (no pain) and 10 is the maximum value (maximum pain).

CONTACTS AND LOCATIONS:
Locations (1):
- Nutrition and Exercise Lab, DSB, University of Padova, Padua, Italy